CLINICAL TRIAL: NCT05679609
Title: Value of Incentive Spirometry in Routine Management of COPD Patients and Its Effect on Diaphragmatic Function
Brief Title: Incentive Spirometry in Routine Management of COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal A. El-Koa, doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6/2022CHES4-1
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: COPD
Keywords: COPD; incentive spirometry; diaphragmatic ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): participants would use incentive spirometry for 2 months together with ordinary medical treatment
  Interventions: Device: incentive spirometry
- group 2 (No Intervention): participants would receive only ordinary medical treatment for 2 months

INTERVENTIONS:
Device: incentive spirometry — It is flow-oriented that has 3 chambers, (600, 900, and 1200 cc/s) and it has a mouthpiece and a ball in each chamber. After a quiet exhalation, each participant was instructed to take slow full inspirations and to keep as long as he can for at least 5 seconds, then he slowly expires. The device is used every hour at least 5 to 10 times in the session during wake time.
  Arms: group 1

SUMMARY:
The incentive spirometer is a device that encourages patients, with visual and other positive feedback, to maximally inflate their lungs and sustain that inflation. However, its efficacy in patients with COPD has been little documented especially in diaphragmatic function. This study tried to assess the role of incentive spirometry on Spirometric functions, Sonographic diaphragmatic function, and the scale of dyspnea in COPD patients with exacerbation and with follow-up of these parameters after 2 months.

DETAILED DESCRIPTION:
Forty COPD patients were admitted with an acute exacerbation and the patients were divided randomly into 2 equal groups: the first used the incentive spirometer together with medical treatment (according to GOLD guidelines) for 2 months and the second received only medical treatment for 2 months. All participants, on admission, underwent assessment of mMRC dyspnea scale, spirometry, arterial blood gases, and diaphragmatic ultrasound. Then, a follow-up of the participants was done after 2 months with the same parameters and a comparison between both groups was done.

ELIGIBILITY:
Inclusion Criteria:

* confirmed cases of COPD according to the criteria GOLD
* age more than 40 years

Exclusion Criteria:

* bad acoustic window by ultrasound
* other chronic respiratory diseases
* lung malignancy
* recent major surgery
* inability to complete or perform the study
* patient refusal

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
assessing the change in baseline diaphragmatic excursion in cm | 2 months
  assessing the change from Baseline diaphragmatic excursion (in cm) using ultrasound to 2 months
assessing the change in baseline percentage of diaphragmatic thickness fraction | 2 months
  assessing the change from baseline percentage of diaphragmatic thickness fraction (%) using ultrasound to 2 months
assessing the change in baseline forced vital capacity percentage of predicted | 2 months
  assessing the change from baseline forced vital capacity percentage of predicted (%) using spirometry to 2 months
assessing the change in baseline forced expiratory volume in 1st second/forced vital capacity percentage (%) | 2 months
  assessing the change from baseline forced expiratory volume in 1st second/forced vital capacity percentage (%) using spirometry to 2 months
assessing the change in baseline peak expiratory flow rate percentage | 2 months
  assessing the change from baseline peak expiratory flow rate percentage (%) using spirometry to 2 months
change in arterial blood gases | 2 months
  assessment the change in baseline PaO2 and PaCO2 (in mmHg) to 2 months
assessing the change in mMRC dysnea scale | 2 months
  assessing the change in the severity of dyspnea by mMRC dysnea scale from baseline to 2 months. It is 5 statements giving grades from 0 to 4 with the higher the degree, the more severe the shortness of breath in patients with COPD

CONTACTS AND LOCATIONS:
Locations (1):
- Amal A. El-Koa, Cairo, Egypt

REFERENCES:
- [Background] GBD Chronic Respiratory Disease Collaborators. Prevalence and attributable health burden of chronic respiratory diseases, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Respir Med. 2020 Jun;8(6):585-596. doi: 10.1016/S2213-2600(20)30105-3. PMID 32526187
- [Background] Scherer TA, Spengler CM, Owassapian D, Imhof E, Boutellier U. Respiratory muscle endurance training in chronic obstructive pulmonary disease: impact on exercise capacity, dyspnea, and quality of life. Am J Respir Crit Care Med. 2000 Nov;162(5):1709-14. doi: 10.1164/ajrccm.162.5.9912026. PMID 11069801
- [Background] Petrovic M, Reiter M, Zipko H, Pohl W, Wanke T. Effects of inspiratory muscle training on dynamic hyperinflation in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:797-805. doi: 10.2147/COPD.S23784. Epub 2012 Nov 30. PMID 23233798
- [Background] Barakat S, Michele G, George P, Nicole V, Guy A. Outpatient pulmonary rehabilitation in patients with chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2008;3(1):155-62. doi: 10.2147/copd.s2126. PMID 18488439
- [Background] Cortopassi F, Castro AA, Porto EF, Colucci M, Fonseca G, Torre-Bouscoulet L, Iamonti V, Jardim JR. Comprehensive exercise training improves ventilatory muscle function and reduces dyspnea perception in patients with COPD. Monaldi Arch Chest Dis. 2009 Sep;71(3):106-12. doi: 10.4081/monaldi.2009.355. PMID 19999956
- [Background] Stock MC, Downs JB, Gauer PK, Alster JM, Imrey PB. Prevention of postoperative pulmonary complications with CPAP, incentive spirometry, and conservative therapy. Chest. 1985 Feb;87(2):151-7. doi: 10.1378/chest.87.2.151. PMID 3881226
- [Background] AARC (American Association for Respiratory Care) clinical practice guideline. Incentive spirometry. Respir Care. 1991 Dec;36(12):1402-5. No abstract available. PMID 10145589
- [Background] Casaburi R, Porszasz J, Burns MR, Carithers ER, Chang RS, Cooper CB. Physiologic benefits of exercise training in rehabilitation of patients with severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 May;155(5):1541-51. doi: 10.1164/ajrccm.155.5.9154855.
- [Background] Darnley GM, Gray AC, McClure SJ, Neary P, Petrie M, McMurray JJ, MacFarlane NG. Effects of resistive breathing on exercise capacity and diaphragm function in patients with ischaemic heart disease. Eur J Heart Fail. 1999 Aug;1(3):297-300. doi: 10.1016/s1388-9842(99)00027-6. PMID 10935679
- [Background] Cheng YY, Lin SY, Hsu CY, Fu PK. Respiratory Muscle Training Can Improve Cognition, Lung Function, and Diaphragmatic Thickness Fraction in Male and Non-Obese Patients with Chronic Obstructive Pulmonary Disease: A Prospective Study. J Pers Med. 2022 Mar 16;12(3):475. doi: 10.3390/jpm12030475. PMID 35330474